CLINICAL TRIAL: NCT07235540
Title: The Use of a Hyperthermia Pelotte to Acquire More Representative Vaginal Temperature Measurements During Deep Hyperthermia Treatments for Gynaecological Cancer; a Comparative Cross-over Study.
Brief Title: More Representative Vaginal Temperature Measurements With a Hyperthermia Pelotte During Hyperthermia Treatments for Gynaecological Cancer.
Acronym: ORIENTATE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. G.H. (Henrike) Westerveld (Other)
Responsible Party: Sponsor-Investigator, Dr. G.H. (Henrike) Westerveld, Dr., Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: NL-010698
Record Dates: First submitted 2025-11-13; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Gynaecologic Cancer
Keywords: Pelotte; Hyperthermia; Probe; Gynaecologic
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Intervention Model Description: The participants will be treated at least two treatments with pelotte and at least two with a standard vaginal probe.
  Based on a sample size calculation, 27 participants need to be included to achieve sufficient statistical power. Additionally, these data will be used to complete the MDR procedure for the pelotte (clinical validation).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other): Participants will be treated with a pelotte in treatment 1,3 and 5
  Interventions: Device: Pelotte
- Group 2 (Other): Participants will be treated with a pelotte in treatment 1,2 and 4
  Interventions: Device: Pelotte

INTERVENTIONS:
Device: Pelotte — The pelotte is a medical device. It is a round rod made of PTFE - polytetrafluoroethylene (figure 3). The top 7 cm has a diameter of 20 mm and the bottom 13 cm has a diameter of 11 mm. One disposable catheter for temperature measurements will be attached to the pelotte with tape. This catheter will be placed ventrally on the pelotte. A thermometer will be placed in this catheter. This thermometer will measure the vaginal temperatures. A condom is then placed over the pelotte and the catheter before insertion into the patient.
  At least two treatment will be with pelotte and at least 2 with a standard vaginal probe.

SUMMARY:
The goal of this comparative, cross over single centre study is to to determine whether the average measured vaginal temperature during hyperthermia treatment is (clinically) significant different with the use of a pelotte than with a standard vaginal probe. in 27 women treated with external beam radiotherapy and deep hyperthermie for gynaecological cancer.. The primary endpoint is measured average vaginal temperatures with pelotte versus a standard vaginal probe.

The secondary endpoints are: reproducibility of catheter placement, patient comfort, inter-fractional spread of the vaginal temperature and the average vaginal temperature at the tip (0 cm) and 2 cm from the tip with pelotte and a standard vaginal probe.

Participants will be treated at least two time with a pelotte and two times with a standard vaginal probe. Participants will be asked to fill in a short questionnaire three times per treatment (before, during and after treatment). A total of 12-15 questionnaires will be completed by the participants over the four to five treatments.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 or older diagnosed with gynaecological cancer
* Indication for EBRT with DHT
* Written informed consent

Exclusion Criteria:

* Any condition potentially interfering with the understanding of the study requirements, informed consent procedure and completion of questionnaires
* If the vaginal lumen is <4 cm.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2028-01-05 (Estimated); Study Completion 2028-01-05 (Estimated)

PRIMARY OUTCOMES:
• Average vaginal temperature during DHT treatments with pelotte and with a standard vaginal probe. | approximately seven weeks from the intake with the radiation oncologist to the last treatment administration
  To compare if the average vaginal measured temperature is significant different with a pelotte versus the standard vaginal probe

SECONDARY OUTCOMES:
Inter-fractional reproducibility of the catheter placement in depth and position with pelotte and with a standard vaginal probe. | Approximately seven weeks from the intake with the radiation oncologist to the last treatment administration
  For each treatment, the free length of the vaginal probe is measured from the outer labia to the probe tip. This distance is subtracted from 293 mm to determine the internal depth of the vaginal probe. In the control room, the depth is determined based on the temperature measurements. If the measured temperature falls below 36 degrees Celsius at a certain point (e.g., 8 cm from the tip), this point is considered the probe depth. These values are then compared to assess whether there is a difference in reproducibility between treatments using the pelotte and treatments using only a vaginal probe.
Inter-fractional variance in measured vaginal temperatures with pelotte and with a standard vaginal probe. | Approximately seven weeks from the intake with the radiation oncologist to the last treatment administration.
Patient-reported comfort with pelotte and with a standard vaginal probe, as assessed using the 'Vragenlijst Hyperthermie Pelotte' questionnaire | Approximately seven weeks from the intake with the radiation oncologist to the last treatment administration.
Average vaginal temperature at the measurement points of the tip (0 cm) and two cm from the tip of the catheter with pelotte and with a standard vaginal probe. | Approximately seven weeks from the intake with the radiation oncologist to the last treatment administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, South Holand, Netherlands

IPD SHARING:
Plan to Share IPD: No